CLINICAL TRIAL: NCT06364644
Title: Understanding and Addressing Risks of Low Socioeconomic Status and Diabetes for Heart Failure (UNLOAD-Heart Failure)
Brief Title: Understanding and Addressing Risks of Low Socioeconomic Status and Diabetes for Heart Failure
Acronym: UNLOAD-HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00336599; 1P50MD017348-01 (NIH)
Record Dates: First submitted 2024-03-27; First posted 2024-04-15 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Type2diabetes; Heart Failure; Obesity
Keywords: Behavioral Intervention; Diabetes; Heart Failure; Exercise; Obesity; Health Equity; Low Socioeconomic Status
MeSH Terms: conditions — Heart Failure; Obesity; Diabetes Mellitus; Motor Activity | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: The design of the study is a randomized 2:1 parallel-arm clinical trial.
Who Masked: Outcomes Assessor
Masking Description: Participants and interventionists will be unblinded, while those assessing outcomes will be blinded to the randomization arm .
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community Champions (Experimental): Participants assigned to the "Community Champions" group will undergo a six-month behavioral intervention. This intervention involves bi-weekly problem-solving training sessions (DECIDE) conducted in groups of 6-10 individuals, along with support from community health workers. Additionally, participants will receive a YMCA membership to exercise with a professional health coach.
  Interventions: Behavioral: Community Champions
- Homegrown Heroes (Active Comparator): Participants assigned to the "Homegrown Heroes" will receive a YMCA membership for exercise and a monthly newsletters for 6 months that include education about diabetes self-management, healthy lifestyle and heart failure prevention .
  Interventions: Behavioral: Homegrown Heroes

INTERVENTIONS:
Behavioral: Community Champions — The UNLOAD-Heart Failure Program intervention includes problem solving training, community health worker support, and exercise support from health coaches at YMCAs.
  Other Names: Multi-level intervention
  Arms: Community Champions
Behavioral: Homegrown Heroes — Monthly newsletters/videos on diabetes self-management, healthy lifestyle and heart failure prevention will be provided, as well as a membership to the local YMCA.
  Other Names: Education plus access to community exercise facility
  Arms: Homegrown Heroes

SUMMARY:
This study aims to determine whether a 6-month multilevel intervention involving problem-solving training, exercise training and support from community health workers is more effective in improving outcomes for individuals with low socioeconomic status, type 2 diabetes, obesity, and early cardiac dysfunction than receiving education and access to a community exercise facility.

DETAILED DESCRIPTION:
This randomized controlled trial employs a 2:1 allocation ratio. The study aims to include 402 individuals from Baltimore City and Hagerstown, Maryland, characterized by low neighborhood and individual socioeconomic status, type 2 diabetes, obesity, and evidence of subclinical heart dysfunction, without a prior clinical diagnosis of heart failure. The 6-month multi-level intervention consists of three key components:

1. Problem Solving - Diabetes Self-Management Training (DECIDE): Participants will engage in a biweekly evidence-based behavioral change program known as DECIDE. This program focuses on problem-solving training, aiding individuals in managing chronic conditions by overcoming obstacles and challenges. It aims to enhance self-care, improve control of metabolic risk factors, and includes tailored education on heart failure prevention.
2. Community Health Worker Support: Participants will receive ongoing support from community health workers as part of the intervention. These workers will conduct telephone and/or home visits at least monthly, offering assistance in following areas:

   * Reinforcing patient education about disease self-management
   * Helping patients access care and addressing barriers to care and treatment
   * Serving as facilitators and navigators to clinical care, social services, and other community resources
   * Providing encouragement and support to engage, activate, and empower patients and their support systems
3. Health Coaching and Partnership with Community Facilities: Participants will engage in supervised aerobic and resistance exercise training at the local Young Men's Christian Associations (YMCAs). The participants will receive instructions on gradually increasing the activity levels throughout the 6-month intervention to achieve physical activity goals (150 minutes of moderate to vigorous exercise per week).

ELIGIBILITY:
Inclusion Criteria:

* Adults from Johns Hopkins Medicine (JHM) who live in Baltimore City and adults from Johns Hopkins Community Physicians (JHCP) Hagerstown or Family Healthcare of Hagerstown who live in Washington County
* Low socioeconomic status (SES) by high Area Deprivation Index (ADI) [>75th percentile for the state of Maryland] plus low income)
* Type 2 diabetes
* Obesity (BMI≥30 kg/m^2)

Exclusion Criteria:

* Age < 30 or >70 years
* Prevalent heart failure
* Uncontrolled glycemia (blood glucose <60 mg/d or ≥ 300 mg/dl or most recent hemoglobin A1c ≥11%)
* Uncontrolled blood pressure (Systolic blood pressure (SBP) ≥160 or diastolic blood pressure (DBP) ≥100 mm Hg, either on or off medications)
* Known coronary artery disease (unless < 50% stenosis by angiography)
* Moderate or severe valvular heart disease
* Serious medical conditions limiting life expectancy or requiring active management
* Inability to participate in moderate intensity physical activity as assessed by the self-report Physical Activity Readiness Questionnaire Plus (PAR-Q+).
* Weight loss of ≥ 5% in the past year or current use of weight loss medications
* Any condition or planned surgery/procedure precluding exercise for ≥ 150 minutes per week
* End stage renal disease
* Current participation in another behavior change program
* Active alcohol or substance abuse disorder
* Already engaging in regular exercise with more than 60 minutes of moderate [3-6 METS] to vigorous [>6 METS] physical activity per week
* Active pregnancy
* Evidence of ischemia, dangerous arrhythmia or other clinical instability on baseline exercise stress test

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Change in fitness as assessed by the 6 minute walk test | Baseline and 6 month follow up
  Total distance walked in the 6 minutes walk test in meters

SECONDARY OUTCOMES:
Change in cardiac biomarker, high-sensitivity cardiac troponin-T (hs-cTnT) | Baseline and 6 month follow up
  Percent change from baseline in hs-cTnT
Change in hemoglobin A1c | Baseline and 6 month follow up
  Absolute change from baseline in hemoglobin A1c
Change in specific problem solving skills as assessed by Health Problem-Solving Scale (HPSS) subscales. | Baseline, 6 month follow up, 12 month follow up
  The following Health Problem-Solving Scale (HPSS) subscales will be assessed: Impulsive/Careless Problem Solving (IPS), Avoidant Problem Solving (APS), Negative Transfer (NTR), Negative Motivation/Orientation (NMO). Subscale scores are calculated by summing the scores for each item within the respective subscales. Higher subscale scores indicate more of that problem-solving characteristic. The score range for each subscale is as follows: IPS (0-32), APS (0-28), NTR (0-44), NMO (0-20). Total score range 0-124.
Changes in self care measures as assessed by Summary of Diabetes Self-Care Activities Scale (SDSCA) | Baseline, 6 month follow up, 12 month follow up
  The Summary of Diabetes Self-Care Activities Scale (SDSCA) is a tool used to measure diabetes self-care activities. 12-items with 5 sub-scales (diet, exercise, home blood glucose testing, foot care, smoking status). The respondent is asked how many days in the past week the behavior was performed (ranges from 0 to 7); The result is an average score between 0 and 7 with higher score indicating better diabetes self-management behavior.
Changes in disease knowledge as assessed by Diabetes and Cardiovascular Disease (CVD) Knowledge Test | Baseline, 6 month follow up, 12 month follow up
  The Diabetes and CVD Knowledge Test comprises 16 items, featuring both multiple-choice and true-or-false questions. This assessment tool gauges individuals' comprehension of diabetes, its impact on health, and optimal strategies for managing the condition. The possible score range is 0-17. A higher score indicates a better understanding of diabetes and cardiovascular disease.
Changes in physical activity as assessed by Modified Physical Activity Questionnaire (MPAQ) | Baseline, 6 month follow up, 12 month follow up
  The MPAQ is a tool used to estimate the frequency in days (number of times per month) and in time (minutes) someone participated in physical activity (e.g. biking, walking, swimming, etc.). Hours per week for all activities are summed to determine activity hours per week averaged over the past year. A higher sum indicates more physical activity. Values can also be weighted by their estimated metabolic cost and expressed as metabolic equivalent (MET) hours per week. Higher METs are associated with better outcomes.
  The MPAQ also assesses inactivity, such as the average number of hours per day spent watching television or being confined to a bed or chair for more than 1 week. A higher average indicates less physical activity.
Change in weight (kgs) | Baseline and 6 month follow-up
  Change from baseline in weight (kgs)
Change in BMI | Baseline and 6 month follow-up
  Change from baseline in BMI (Kg/m^2).
Change in hip and waist circumference (centimeters) | Baseline and 6 month follow up
  Change from baseline in hip and waist circumference (centimeters)
Change in Metabolic Syndrome Severity Z score | Baseline and 6 month follow up
  Metabolic Syndrome Severity (MetS) Z score calculates an individual's metabolic syndrome severity score by examining five key markers: waist circumference, blood pressure, triglycerides, HDL, and fasting glucose. Score typically ranges from -5 to 5. Higher scores indicate greater metabolic syndrome severity.
Change in self-management as assessed by the Patient Activation Measure (PAM-13). | Baseline, 6 month follow up,12 month follow up
  The Patient Activation Measure is a 13-item survey that will assess an individual's knowledge, skills and confidence to managing one's health and healthcare. The PAM scores is calculated and then transformed to a scale with a range from 0-100. A higher PAM score indicates higher patient activation. The score can also be converted into four activation levels: 1 - not believing activation important, 2 - lack of knowledge and confidence to take action, 3 - beginning to take action, 4 - taking action.
Change in quality of life and overall health and well-being as assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health 10 | Baseline, 6 month follow up,12 month follow up
  The PROMIS Global Health 10 survey comprises 10 items designed to evaluate both physical and mental health status. Scores are aggregated separately for physical and mental health, each ranging from 4 - 20. Higher scores in both categories indicate better outcomes.
Change in blood pressure (systolic and diastolic (mmHg)) | Baseline and 6 month follow up
  changes in blood pressure from baseline
Change in cardiac biomarker, gal-3 | Baseline and 6 month follow up
  Percent change from baseline in gal-3
Change in cardiac biomarkers, NT-proBNP | Baseline and 6 month follow up
  Percent change from baseline in NT-proBNP
Change in post-walk Borg dyspnea scale | Baseline and 6 month follow up
  Changes in post-walk Borg dyspnea scale which ranges from 0 ("no shortness of breath") to 10 ("worst possible shortness of breath"); higher score worse breathing difficulty. Measured in a subset of the population.
Change in cardiorespiratory fitness as assessed by peak oxygen uptake (V02 peak) | Baseline and 6 month follow up
  Change in peak oxygen uptake (VO2 peak) as assessed by a cardiopulmonary fitness test in a subset of the population.

CONTACTS AND LOCATIONS:
Overall Officials: Chiadi Ndumele, MD, PhD, Principal Investigator — Johns Hopkins School of Medicine
Locations (2):
- United States (2):
  - Johns Hopkins Center for Health Equity, Baltimore, Maryland
  - Johns Hopkins University Comstock Center, Hagerstown, Maryland

IPD SHARING:
Plan to Share IPD: No